CLINICAL TRIAL: NCT04269148
Title: Validity and Reliability of the Turkish Version of the McMaster University Head and Neck Radiotherapy Questionnaire
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Izmir Bakircay University (Other)
Collaborators: Gazi University (Other)
Responsible Party: Principal Investigator, Kadirhan Ozdemir, PT, PhD., Head of Geriatric Rehabilitation Department, Izmir Bakircay University
Other Study IDs: 2018-147
Record Dates: First submitted 2020-02-08; First posted 2020-02-13 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Quality of Life; Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Head and Neck Cancer patients: Turkish patients diagnosed with head and neck cancer
  Interventions: Other: Measurement of Quality of Life

INTERVENTIONS:
Other: Measurement of Quality of Life — Quality of life will be measured using McMaster University Head and Neck Radiotherapy Questionnaire and The Functional Assessment of Cancer Therapy - Head and Neck Cancer Version 4

SUMMARY:
More than half of the patients with head and neck cancer are locally advanced patients. Radiotherapy is the primary treatment option for many patients with stage III and stage IV diagnosed with head and neck cancer. Radiation often causes tissue reactions by increasing local symptoms of the tumor and adding new symptoms to them. The acute effects of radiation are pain and burns associated with mucosal irritations and skin irritations, the root smell of the necrotic tumor and damaged normal tissues, dry skin, skin irritation, pain and dryness of mucosal membranes, decreased appetite, loss of chewing and swallowing skills, and hoarseness. The aim of this study is to make the validity, reliability and cultural adaptation of McMaster University Head and Neck Radiotherapy Inventory in Turkish.

DETAILED DESCRIPTION:
Although there are various surveys in the literature that evaluate the quality of life of head and neck cancer patients, apart from the "McMaster University Head and Neck Radiotherapy Questionnaire", there is no other questionnaire designed specifically for local advanced stage III and stage IV head and neck cancer and treatment of specific morbidity at a certain time. Patients in these stages often have difficulties in oral communication, nutritional disorders and loss of chewing and swallowing skills leading to dehydration, bad mouth odors, appearance problems affecting social and family life, and often significant morbidity including severe pain symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily accepting to participate in the study
* Patients whose native language is Turkish
* Undergoing or receiving radiotherapy treatment
* At least 3 weeks have passed since the beginning of radiotherapy

Exclusion Criteria:

* The patient does not have sufficient functions of bone marrow, liver and kidney
* To have scored less than 70 from Karnofsky Performance Scale

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Turkish patients diagnosed with head and neck patients
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2020-03-13 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
McMaster University Head and Neck Radiotherapy Questionnaire | At baseline
  McMaster University Head and Neck Radiotherapy Questionnaire: This questionnaire includes 22 questions covering signs and symptoms related to 6 categories: oral cavity, throat, skin, digestive system, energy and psychosocial. n each category, there are at least 3 questions related to that category. There are 7 possible answer options in each question using Likert scale. High scores obtained according to the scoring system used indicate low toxicity. The final score of the survey is expressed as the average of the scores from 22 questions. In addition, the independent scores of each category are the average of the scores from the questions belonging to that category [1].

SECONDARY OUTCOMES:
The Functional Assessment of Cancer Therapy - Head and Neck Cancer Version 4 | At baseline
  This scale consists of 5 categories that evaluate physical (7 items), social (7 items), emotional (6 items), functional status (7 items) and a subscale consisting of 11 questions specifically developed for head and neck cancer. In this assessment consisting of 38 items in total, each field can be scored among themselves and a total score is also calculated. The increase in the total score shows that the quality of life is higher. Each item is scored by patients with a Likert type classification ranging from 0 (none) to 4 (too many).

CONTACTS AND LOCATIONS:
Locations (1):
- Kadirhan Ozdemir, Izmir, Turkey (Türkiye)

REFERENCES:
- [Background] Browman GP, Levine MN, Hodson DI, Sathya J, Russell R, Skingley P, Cripps C, Eapen L, Girard A. The Head and Neck Radiotherapy Questionnaire: a morbidity/quality-of-life instrument for clinical trials of radiation therapy in locally advanced head and neck cancer. J Clin Oncol. 1993 May;11(5):863-72. doi: 10.1200/JCO.1993.11.5.863. PMID 8487051
- [Background] List MA, D'Antonio LL, Cella DF, Siston A, Mumby P, Haraf D, Vokes E. The Performance Status Scale for Head and Neck Cancer Patients and the Functional Assessment of Cancer Therapy-Head and Neck Scale. A study of utility and validity. Cancer. 1996 Jun 1;77(11):2294-301. doi: 10.1002/(SICI)1097-0142(19960601)77:113.0.CO;2-S. PMID 8635098
- [Background] Webster K, Cella D, Yost K. The Functional Assessment of Chronic Illness Therapy (FACIT) Measurement System: properties, applications, and interpretation. Health Qual Life Outcomes. 2003 Dec 16;1:79. doi: 10.1186/1477-7525-1-79. PMID 14678568